CLINICAL TRIAL: NCT07150975
Title: A Multicenter, Randomized, Open-Label, Parallel-Group Phase III Clinical Study Comparing the Efficacy and Safety of GZR18 Injection and Semaglutide(Wegovy®) in Adult Obese or Overweight Subjects
Brief Title: Phase III Clinical Study Comparing the Efficacy and Safety of GZR18 Injection and Semaglutide (Wegovy®) in Adult Obese or Overweight Subjects
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gan & Lee Pharmaceuticals. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZR18-BWM-302
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Obesity/Overweight in Adult
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GZR18 Dose Level 1 (Experimental)
  Interventions: Drug: GZR18
- GZR18 Dose Level 2 (Experimental)
  Interventions: Drug: GZR18
- Semaglutide(Wegovy® )2.4 mg (Active Comparator)
  Interventions: Drug: Semaglutide(Wegovy® )

INTERVENTIONS:
Drug: GZR18 — Administered SC
  Arms: GZR18 Dose Level 1; GZR18 Dose Level 2
Drug: Semaglutide(Wegovy® ) — Administered SC
  Arms: Semaglutide(Wegovy® )2.4 mg

SUMMARY:
This study is a multicenter, randomized, open-label, parallel-group phase III clinical trial comparing the efficacy and safety of GZR18 Injection and semaglutide (Wegovy®) in adult obese or overweight subjects, aiming to evaluate the efficacy and safety of GZR18 Injection in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years old (based on the date of signing the informed consent form), male or female.
2. For subjects not diagnosed with type 2 diabetes at screening, the following criteria must be met:

   At screening and Visit 2 (before randomization), the subject must be either obese (BMI ≥ 28 kg/m²) or overweight (24 kg/m² ≤ BMI < 28 kg/m²), and concurrently present with at least one of the following conditions:
   * Comorbidity of one or more of the following: hyperglycemia (see Appendix 1 for definition), hypertension, dyslipidemia (see Appendix 2 for definition), or fatty liver; ②Weight-bearing joint pain;

     * Weight-related obstructive sleep apnea syndrome.
3. For subjects with type 2 diabetes at screening, the following criteria must be met simultaneously:

   Body mass index (BMI) ≥ 24 kg/m² at both screening and Visit 2 (before randomization); A confirmed diagnosis of type 2 diabetes for at least 90 days at screening, in accordance with the World Health Organization (WHO) 1999 diabetes diagnostic criteria and the 2011 supplementary diagnostic criteria (HbA1c-based diagnosis is recommended); Within 90 days prior to screening: ① Management through diet and exercise alone, with no use of any antidiabetic medications; or ② Treatment of type 2 diabetes with a stable dose of metformin monotherapy, where the metformin dose is ≥ 1500 mg/day or the maximum tolerated dose (< 1500 mg/day but ≥ 1000 mg/day); or ③ Treatment of type 2 diabetes with a stable dose of metformin (≥ 1500 mg/day or the maximum tolerated dose (< 1500 mg/day but ≥ 1000 mg/day)) combined with a stable dose of sodium-glucose cotransporter 2 inhibitor (SGLT2i); Glycated hemoglobin (HbA1c) measured by the central laboratory at screening is 7.0-10.5% (inclusive of both endpoints); Fasting plasma glucose measured by the central laboratory at screening is < 15 mmol/L.
4. Prior to screening, the subject has been managed by diet and exercise alone for at least 12 weeks, and the body weight change has been < 5% within the past 12 weeks (based on self-report).
5. Subjects of childbearing potential must have no childbearing plans from the time of signing the informed consent form to 8 weeks after the last dose, and voluntarily adopt effective contraceptive measures, with no plans for sperm/egg donation. Females of childbearing potential must not be breastfeeding, and the pregnancy test results must be negative at both screening and Visit 2 (before randomization).
6. The subject must be able to understand the procedures and methods of this study, be willing and able to maintain a regular diet and exercise lifestyle during the study period, be willing and able to receive subcutaneous injection of the investigational product, and voluntarily sign the informed consent form.

   -

Exclusion Criteria:

1. For subjects without type 2 diabetes at screening, the following situations are excluded:

   * Fasting plasma glucose ≥ 7.0 mmol/L or glycated hemoglobin (HbA1c) ≥ 6.5% as measured by the central laboratory at screening.

     * Diagnosis of any type of diabetes (excluding gestational diabetes) prior to screening.

       * Use of glucagon-like peptide-1 receptor (GLP-1R) agonists or drugs with a GLP-1R agonist mechanism of action (e.g., GLP-1R/glucagon receptor (GCGR) agonists, glucose-dependent insulinotropic polypeptide receptor (GIPR)/GLP-1R agonists, or GIPR/GLP-1R/GCGR agonists, etc.) prior to screening.
2. For subjects with type 2 diabetes at screening, the following situations are excluded:

   * Use of glucagon-like peptide-1 receptor (GLP-1R) agonists or drugs with a GLP-1R agonist mechanism of action (e.g., GLP-1R/glucagon receptor (GCGR) agonists, glucose-dependent insulinotropic polypeptide receptor (GIPR)/GLP-1R agonists, or GIPR/GLP-1R/GCGR agonists, etc.) within 180 days prior to screening; or a history of poor blood glucose control efficacy or intolerance to the above-mentioned drugs (as assessed by the investigator).

     * A history of diabetic ketoacidosis, lactic acidosis, or hyperosmolar hyperglycemic state within 180 days prior to screening.

       * Presence of severe chronic diabetic complications at screening (e.g., proliferative retinopathy or macular edema, painful diabetic neuropathy, intermittent claudication, or diabetic foot).

         * A history of refractory or complicated urinary tract infections/genital infections within 6 months prior to screening.
3. Subjects with known or suspected allergies to glucagon-like peptide-1 (GLP-1) receptor agonists or their excipients.
4. A history of substance abuse prior to screening.
5. A history of alcohol abuse within 180 days prior to screening, defined as an average weekly alcohol intake exceeding 14 units (for males)/7 units (for females) (1 standard unit is equivalent to 360 mL of beer, 150 mL of wine with 12% alcohol content, or 45 mL of spirits with 40% alcohol content).
6. Presence of limb deformities or disabilities that affect height measurement.
7. Previous receipt of bariatric surgery prior to screening, or planned receipt of bariatric surgery during the study period (exceptions include acupuncture for weight loss, liposuction, or abdominal liposuction performed more than 1 year prior to screening; and removal (or expulsion) of intragastric balloons more than 1 year prior to screening).
8. Obesity caused by secondary diseases or medications, including: elevated cortisol (e.g., Cushing's syndrome), obesity due to pituitary or hypothalamic damage, etc.
9. A history of severe hypoglycemia or grade 3 hypoglycemia within 180 days prior to screening.
10. A personal history or relevant family history of medullary thyroid carcinoma, multiple endocrine neoplasia (MEN) type 2A or 2B prior to screening; or a history of malignant tumors within the past 5 years (excluding cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix).
11. The investigator deems that the subject has any other factors that may affect the evaluation of efficacy or safety in this study, making them unsuitable for participation.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline after 52 weeks (W) of treatment. | From Week 0 to Week 52

SECONDARY OUTCOMES:
Efficacy Outcome Measure :Percentage of subjects with body weight reduction ≥ 5% from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Percentage of subjects with body weight reduction ≥ 10% from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Percentage of subjects with body weight reduction ≥ 15% from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Percentage of subjects with body weight reduction ≥ 20% from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Percentage of subjects with body weight reduction ≥ 25% from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Changes in body weight from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Changes in body mass index (BMI) from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Changes in waist circumference from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Changes from baseline in glycated hemoglobin (HbA1c) | From Week 0 to Week 52
Efficacy Outcome Measure :Changes from baseline in fasting plasma glucose | From Week 0 to Week 52
Efficacy Outcome Measure :Changes from baseline in fasting insulin | From Week 0 to Week 52
Efficacy Outcome Measure :Changes insystolic blood pressure from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Changes in diastolic blood pressure from baseline | From Week 0 to Week 52
Efficacy Outcome Measure :Changes from baseline in total cholesterol (TC) | From Week 0 to Week 52
Efficacy Outcome Measure :Changes from baseline in low-density lipoprotein cholesterol (LDL-C) | From Week 0 to Week 52
Efficacy Outcome Measure :Changes from baseline in high-density lipoprotein cholesterol (HDL-C) | From Week 0 to Week 52
Efficacy Outcome Measure :Changes from baseline in triglycerides (TG) | From Week 0 to Week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing, Beijing, China